CLINICAL TRIAL: NCT02491281
Title: A Randomized, Placebo Controlled, Double-blind First-in-human Single Ascending Dose Study of LNA043 in Primary Osteoarthritis Patients Scheduled for Total Knee Replacement
Brief Title: First-in-human Single Ascending Dose Study of LNA043 in Patients Scheduled for Total Knee Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: CLNA043X2101
Record Dates: First submitted 2015-06-23; First posted 2015-07-08 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2018-08

CONDITIONS: Primary Osteoarthritis Patients Scheduled for Total Knee Replacement Surgery
Keywords: Primary Osteoarthritis, Total Knee Replacement, cartilage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNA043 (Experimental): LNA043 given intra-articularly
  Interventions: Drug: LNA043
- Placebo (Placebo Comparator): Placebo given intra-articularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNA043 — ascending single dose on Day 1; 1 to 4 week(s) prior total knee replacement surgery
  Arms: LNA043
Drug: Placebo — ascending single dose on Day 1; 1 to 4 week(s) prior total knee replacement surgery
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and tolerability of ascending single doses of LNA043 given intra-articularly into the human knee joint prior to its removal at total knee replacement surgery. In addition, this will help to establish the presence of LNA043 within the articular cartilage, assess pharmacokinetics and immunogenicity, and will allow exploration of biomarkers of hyaline cartilage repair.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients age 50 to 75 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening
* Patients diagnosed with primary osteoarthritis of the knee assessed locally for whom a total knee replacement is planned
* General health status acceptable for total knee replacement surgery in the opinion of the investigator
* Stable medications within 3 months prior to enrollment (such as appropriate pain medication, antibiotics prophylaxis) and standard of care

Key Exclusion Criteria:

* Presence of inflammatory arthropathy (including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout), active acute or chronic infection, or systemic cartilage disorder
* Prior cartilage repair surgery, e.g. microfracture, autologous cartilage implantation (ACI) or else, at the same knee
* Any surgical therapy or local treatment i.a. into the knee (viscosupplementation) to the knee within 2 months prior to enrollment
* BMI > 40; presence of uncontrolled diabetes or hyperthyroidism
* Large effusion in the knee to be replaced, more than (>)1 cm fluid in the suprapatellar space at the midline
* Corticosteroid use by any route except topical and nasal in the 3 months prior to enrollment
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Safety endpoints (including number of adverse events CTC-AE, physical exam, vital signs, ECG, safety laboratory and pain measured using KOOS) | Up to and including 7 days post-dose
  Safety and tolerability of LNA043 after one intra-articular injection into the knee of osteoarthritis patients scheduled for total knee replacement

SECONDARY OUTCOMES:
Immunohistochemical staining for LNA043 in knee cartilage | 1 up to 4 weeks post-dose
  Joint presence and persistence of LNA043 within the cartilage of the knee
Concentration of LNA043 in serum and synovial fluid | Pre-dose, Day 1, Day 4, Day 8, and Day 36
  LNA043 pharmacokinetics in serum and concentration in synovial fluid to determine local and systemic exposure
Concentration of ANGPTL in serum and synovial fluid | Pre-dose, Day 1, Day 4, Day 8, and Day 36
  ANGPTL levels in serum and the synovial fluid
Presence of anti-LNA043 | Pre-dose, Day 8, and Day 36
  Immunogenicity in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gerwin N, Scotti C, Halleux C, Fornaro M, Elliott J, Zhang Y, Johnson K, Shi J, Walter S, Li Y, Jacobi C, Laplanche N, Belaud M, Paul J, Glowacki G, Peters T, Wharton KA Jr, Vostiar I, Polus F, Kramer I, Guth S, Seroutou A, Choudhury S, Laurent D, Gimbel J, Goldhahn J, Schieker M, Brachat S, Roubenoff R, Kneissel M. Angiopoietin-like 3-derivative LNA043 for cartilage regeneration in osteoarthritis: a randomized phase 1 trial. Nat Med. 2022 Dec;28(12):2633-2645. doi: 10.1038/s41591-022-02059-9. Epub 2022 Dec 1. PMID 36456835
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=454
- See also: Results for CLNA043X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17358